CLINICAL TRIAL: NCT01367626
Title: A Single Dose, 2-Period, 2-Treatment 2-Way Crossover Bioequivalency Study of Letrozole Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Letrozole 2.5 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LETR-T25-PVFD-1
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole (Active Comparator): 2.5 mg tablet
  Interventions: Drug: letrozole
- Fermara (Active Comparator): 2.5 mg tablet
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — 2.5 mg tablet
  Other Names: Femara
  Arms: Fermara
Drug: letrozole — 2.5 mg tablet
  Other Names: Femara
  Arms: letrozole

SUMMARY:
The objective of this study was to prove the bioequivalence of Letrozole Tablet under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

- No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to letrozole or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Copa, PharmD, Principal Investigator — PRAC Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States